CLINICAL TRIAL: NCT03494790
Title: Markers of Inflammation and Metabolism in the ER
Acronym: MIMER
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Johanna Hastbacka, MD,PhD, University of Helsinki
Other Study IDs: HelsinkiU1423/2017
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2020-02

CONDITIONS: Acute Infection; Sepsis
Keywords: MMP; Matrix metalloproteinase; Metabolomics; FGF-21; Quick SOFA; Infection; Triage
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum sample 10ml Plasma lactate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Adult patients with suspected or confirmed infection and who will be sampled for blood culture will be recruited. Blood samples are collected for the analysis of matrix metalloproteinases (MMP) and their inhibitors. We also aim to analyse metabolic changes and use the samples for analysis of blood lactate, metabolomics, and fibroblast growth factor 21 (FGF-21) as well. The primary aim of the study is to test the performance of MMP-8 in finding severely ill patients who will need treatment in high dependency unit or intensive care. The secondary aim is to study the metabolic changes in acutely ill patients with infection.

DETAILED DESCRIPTION:
Adult patients with suspected or confirmed infection and who will be sampled for blood culture (a surrogate for suspected severe infection) will be recruited from three large emergency departments in a University hospital. Two blood samples will be collected: one for the analysis of matrix metalloproteinases, their inhibitor tissue inhibitor of metalloproteinase-1 (TIMP-1), FGF-21 and metabolomic analyses. Another blood sample is for the analysis of blood lactate. Clinical data will be collected to calculate quick SOFA (qSOFA), in order to test whether lactate and/or MMP-8 will improve the prognostic model if they are added to qSOFA. The primary outcome measure is the number of days alive without the need for ICU or high dependency unit treatment. The ability of MMP-8 to discriminate severe infection from uneventful course of the disease will be studied. The secondary aim is to study the metabolic changes in acutely ill patients with infection and compare these variables between survivors and non-survivors. The planned number of patients recruited is 924. During this study the feasibility of a bedside rapid analysis of MMP-8 will be tested in 30 patients and the results obtained using the rapid analyser compared with laboratory results obtained using ELISA.

ELIGIBILITY:
Inclusion Criteria:

Age 18 or more Suspected or confirmed infection Admitted to any of the three emergency departments of university hospital Decision of blood culture

Exclusion Criteria:

Age <18 Cancer with metastases Decision of treatment limitation probable or made Consent not obtainable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients that are admitted to the participating emergency departments, with suspected or confirmed acute infection. A decision of taking a blood culture sample is a surrogate for suspected severe infection.
Sampling Method: Non-Probability Sample
Enrollment: 955 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Days alive without intensive care or high dependency unit treatment | 2 weeks from study admission
  Accounts for patients who survive and need no ICU or high dependency care for the primary infection.

SECONDARY OUTCOMES:
30 day mortality | 30 days
  Number of patients who die within 30 days of admission
90 day mortality | 90 days
  Number of patients who die within 90 days aof admission

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided